CLINICAL TRIAL: NCT00390130
Title: Does the Order in Which Vaccines Are Administered Affect Pain Response? A Randomized, Double-blind, Clinical Trial of Pentacel vs. Prevnar
Brief Title: Does the Order in Which Vaccines Are Administered Affect Pain Response?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Moshe Ipp, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000009089
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Pain
Keywords: Vaccination; Pediatrics; Pain
MeSH Terms: conditions — Pain | interventions — pentacel; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pentacel (Active Comparator): The subjects in this arm will be vaccinated with Pentacel
  Interventions: Drug: Pentacel (DPTaP+Hib)
- Prevnar (Active Comparator): The subjects in this arm will be vaccinated with Prevnar
  Interventions: Drug: Prevnar (conjugated pneumococcal vaccine)

INTERVENTIONS:
Drug: Pentacel (DPTaP+Hib)
  Arms: Pentacel
Drug: Prevnar (conjugated pneumococcal vaccine)
  Arms: Prevnar

SUMMARY:
The objective of this study is to determine whether there should be a predetermined sequence recommended for administering these two vaccines, with the less painful vaccine being given first.

DETAILED DESCRIPTION:
Childhood vaccination is one of the most effective public health measures worldwide, with few serious adverse effects reported. However, pain on vaccination continues to be a frequent occurrence and is the most common cause of childhood iatrogenic pain. In a recent study of paediatricians in the USA, more than ninety percent reported at least one parental vaccine refusal in the past year. The most common concerns cited by parents were short-term reactions and pain from multiple injections.

One of the factors responsible for vaccination pain is the vaccine material itself. Even the same vaccine, when made by different pharmaceutical companies may produce different pain responses. Anecdotal reports from doctors and nurses indicate that Pentacel (DPTaP+Hib) is a relatively painless vaccine to administer whereas Prevnar (conjugated pneumococcal vaccine) causes significant pain on injection and severe distress to the infant being vaccinated. For this reason, many vaccinators administer Pentacel [DPT] prior to Prevnar [PCV] when providing both vaccines in one visit. However, the difference in infant pain responses has not been documented. Although it has been shown that very early pain events affect infants' later experience of pain, it has not been demonstrated that the sequence in which vaccines are administered affects pain response. This study will assess whether there should be a predetermined sequence recommended for administering these two vaccines, with the less painful vaccine (Pentacel) being given first.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant
* 2 - 6 months of age
* receiving primary DPT and PCV vaccinations

Exclusion Criteria:

* chronic illness
* immune deficiency
* immunosuppression
* a history of allergy to DPT or PCV or any of its components
* fever
* any acute illness that prevents the administration of the vaccine

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
pain response to vaccination with Prevnar and Pentacel, as measured by The Modified Behavioral Pain Scale (MBPS) and the Visual Analogue Scale (VAS) | Immediately after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Ipp, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Ipp M, Parkin PC, Lear N, Goldbach M, Taddio A. Order of vaccine injection and infant pain response. Arch Pediatr Adolesc Med. 2009 May;163(5):469-72. doi: 10.1001/archpediatrics.2009.35. PMID 19414694